CLINICAL TRIAL: NCT06586047
Title: Evaluation of PSMA Expression in Triple Negative Breast Cancer Patients Using 18 F-DCFPyL-PET/CT
Brief Title: Breast Cancer PSMA PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Shariftabrizi (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ahmad Shariftabrizi, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202306462
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast cancer, PSMA expression, PET imaging
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET Imaging (Experimental): Triple negative breast cancer patients will undergo FDG PET/CT and Pyl PET/Ct
  Interventions: Diagnostic Test: PET imaging

INTERVENTIONS:
Diagnostic Test: PET imaging — Imaging with FDG PET/CT and Pyl PET/CT

SUMMARY:
The purpose of this research is to determine the expression of Prostate Specific Membrane Antigen(PSMA) in metastatic Triple Negative Breast Cancer (TNBC) patients using Fludeoxyglucose F18 (FDG) PET/CT as the gold standard. The investigators hypothesize that most lesions in metastatic TNBC are PSMA-avid; and thus PSMA-based radionuclide therapy can be a valid treatment option for TNBC, and clinical trials can be designed for this purpose. Thirty metastatic TNBC patients will be enrolled and will be on the study for maximum of 4 weeks.

DETAILED DESCRIPTION:
Prostate Specific Membrane Antigen (PSMA) is not only expressed in prostate cancer and its metastases, but also it is expressed on the neovasculature of many other solid tumors including gastric, lung, adrenal, bladder and renal cell carcinomas. Also, there is evidence that breast carcinomas express PSMA, although this has not been specifically studied in the metastatic TNBC.

The study involves a total of 2 visits and on each visit, patients will undergo a PET imaging. Each patient will first undergo an (FDG) PET/CT and then in few days will undergo an 18F-DCFPyL-PET/CT. The PET scanner is a large machine with a hollow tube that will be used to see how F18 FDG is taken up into the tumor and other tissues. The patients will be asked to lie on the back on a special table that slides into the tube. The sides of the tube will be close to the body. At the first visit patients will be in this scanner for approximately 20 minutes.

The study will evaluate the expression of PSMA via 18 F-DCFPyL-PET/CT in metastatic TNBC patients and compare it with lesion detection rate of FDG PET/CT. PSMA-avid lesions will be detected using the novel agent 18 F-DCFPyL and concordance rate with FDG-avid lesions will be calculated. The standardized uptake values (SUV) of each lesion on both FDG PET/CT and 18F-DCFPyL-PET/CT will be compared to find a correlation between tumor aggressiveness (lesion SUV on FDG PET/CT) and tumor angiogenesis (lesion SUV on 18 F-DCFPyL-PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Female >= 18 years of age
* Patients in distantly metastatic TNBC based on the initial diagnosis biopsy.
* Patient should have FDG positive metastatic lesions on the initial PET/CT scan performed in this study to be further included.

Exclusion Criteria:

* Patients with known active other malignancy.
* Unable to tolerate PET/CT procedure.
* Pregnant or breastfeeding.
* Patients with any medical condition that might compromise the safety of subject during PET acquisitions.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Lesion detection sensitivity analysis | 4 weeks
  Comparing the sensitivity of 18 F-DCFPyL-PET/CT and FDG PET/CT in metastatic lesion detection in triple-negative breast cancer patients.

SECONDARY OUTCOMES:
Quantitative radiotracer uptake analysis | 4 weeks
  To quantitively compare the SUVs in each lesion on 18 F-DCFPyL-PET/CT and FDG PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Healthcare, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided